CLINICAL TRIAL: NCT03841721
Title: Pharmacokinetics/Pharmacodynamics of Oral Linezolid 300 mg/Day in Healthy Volunteers
Brief Title: Linezolid in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Sutep Jaruratanasirikul, Department of Medicine, Faculty of Medicine, Prince of Songkla University, Prince of Songkla University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Linezolid 61087141
Record Dates: First submitted 2019-02-13; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Healthy
Keywords: pharmacokinetic; linezolid; healthy volunteers
MeSH Terms: interventions — Linezolid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- linezolid 300 mg (Experimental)
  Interventions: Drug: Linezolid oral tablet 300 mg/day for 5 day

INTERVENTIONS:
Drug: Linezolid oral tablet 300 mg/day for 5 day — Linezolid oral tablet 300 mg/day for 5 day and blood sample were obtained by direct venipuncture at 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hour after drug administration in day 5

SUMMARY:
Linezolid is the first synthetic antibiotic of oxazolidinone group that can inhibit bacterial protein synthesis. Previous studies have found that linezolid was an effective treatment for multidrug-resistant (MDR) and extensively drug-resistant (XDR) tuberculosis (TB). In addition, the current dosage recommendation (1,200 mg/day) occasionally resulted in serious adverse events including bone marrow suppression and peripheral neuropathy.

The objective study were determine the pharmacokinetics of oral linezolid 300 mg /day in healthy volunteers. This study conducted in six healthy volunteers. All subject received an oral linezolid 300 mg/day by directly observed treatment (DOT) at the same time each day for 5 days. Blood samples were collected on day 5 at 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 and 24 h post dosing. The separated plasma samples were evaluated by ultra-performance liquid chromatography (UPLC). All pharmacokinetic parameters were calculated.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 - 40
* BMI 19 - 24 kg/m2
* normal CLcr
* normal liver function

Exclusion Criteria:

* Subject who pregnant
* Subject who have documented hypersensitivity to linezolid

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Concentration of linezolid in plasma | 24 hour after the linezolid dose
  Individual concentration of linezolid in plasma

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Clinical Pharmacology, Department of Medicine, Faculty of Medicine, Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand